CLINICAL TRIAL: NCT02380807
Title: Effects of Dry Needling on Posture, Spinal Mobility and Trigger Points on Spinal Muscles in Patients With Fibromyalgia Syndrome.
Brief Title: Effects of Dry Needling on Spinal Mobility and Trigger Points in Patients With Fibromyalgia Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UAL- 423
Record Dates: First submitted 2015-02-28; First posted 2015-03-05 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Fibromyalgia; Back Pain
Keywords: Paraspinal Muscles; Trigger Points; Randomized Controlled Trial; Mobility Limitation
MeSH Terms: conditions — Fibromyalgia; Back Pain; Mobility Limitation | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling Therapy (Experimental): Dry Needly Therapy will be assesses in trigger points on latissimus dorsi, iliocostalis muscle, multifidus muscles, and quadratus lumbourum muscle.
  Interventions: Device: Dry Needling
- Cross Tape Therapy (Active Comparator): Cross Tape is a grid-shaped bandage easy aplicacionen different parts of the body that regulates the tension.
  Interventions: Other: Cross Tape Therapy

INTERVENTIONS:
Device: Dry Needling — Dry needling is the use of either solid filiform needles or hollow-core hypodermic needles for therapy of muscle pain, sometimes also known as intramuscular stimulation (IMS). Although dry needling originally utilized only hypodermic needles due to the concern that solid filiform needles had neither the strength or tactile feedback that hypodermic needles provided and that the solid filiform needle could be deflected by "dense contraction knots".
  Arms: Dry Needling Therapy
Other: Cross Tape Therapy — The tape consists of cross bands or strips mesh cross, nonelastic and without any medication, forming a grid-shaped patch. The cross tape will be applied on trigger points.
  Arms: Cross Tape Therapy

SUMMARY:
This study evaluates the effect of Dry Needling on Spinal Mobility and Trigger Points in Patients with Fibromyalgia Syndrome.

DETAILED DESCRIPTION:
Dry Needling is a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points, muscular, and connective tissues for the management of neuromusculoskeletal pain and movement impairments. Dry needling (DN) is a technique used to treat dysfunctions in skeletal muscle, fascia, and connective tissue, and, diminish persistent peripheral nociceptive input, and reduce or restore impairments of body structure and function leading to improved activity and participation.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome diagnosis.
* Aged from 18 to 65 years.
* No regular physical activity.
* Limitation of usual activities due to pain on at least 1 day in the previous 30 days.
* Agreement to attend evening therapy sessions.

Exclusion Criteria:

* Severe physical disability.
* Comorbid conditions (eg, morbid obesity, inflammatory diseases, irritable bowel syndrome, interstitial cystitis).
* Uncontrolled endocrine disorders (eg, hyperthyroidism or hypothyroidism, diabetes).
* Malignancy.
* Psychiatric.
* Illnesses (eg, schizophrenia or substance abuse).
* Medication usage other than as-needed analgesics (excluding long-term narcotics).
* History of surgery.
* History of whiplash injury.
* Presence of a score >9 points in the Beck Depression Inventory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | up to Four Weeks
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain.

SECONDARY OUTCOMES:
Number of participants with Trigger Points | up to Four Weeks
  Dry Needly Therapy will be assesses in trigger points on trapezius muscle, supraspinatus muscle, infraspinatus muscle, latissimus dorsi, iliocostalis muscle, multifidus muscles, and quadratus lumbourum muscle.
Posture and Spinal Mobility | up to Four Weeks
  Spinal Mouse is a device that, combined with a computer program (PC), assesses the curvatures of the vertebral column without applying harmful radiation. Spinal Mouse checks: spine alignment, measuring segmental and global angles in the sagittal and frontal planes; posture and spinal mobility; and spine functions and performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity of Almería, Almería, Almería, Spain

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Arnold LM, Clauw DJ, McCarberg BH; FibroCollaborative. Improving the recognition and diagnosis of fibromyalgia. Mayo Clin Proc. 2011 May;86(5):457-64. doi: 10.4065/mcp.2010.0738. PMID 21531887
- [Background] Goldenberg DL. Fibromyalgia syndrome: an emerging but controversial condition. JAMA. 2014 Apr 16;311(15):1570. doi: 10.1001/jama.2013.279453. No abstract available. PMID 24737378
- [Background] Mas AJ, Carmona L, Valverde M, Ribas B; EPISER Study Group. Prevalence and impact of fibromyalgia on function and quality of life in individuals from the general population: results from a nationwide study in Spain. Clin Exp Rheumatol. 2008 Jul-Aug;26(4):519-26. PMID 18799079
- [Background] Branco JC, Bannwarth B, Failde I, Abello Carbonell J, Blotman F, Spaeth M, Saraiva F, Nacci F, Thomas E, Caubere JP, Le Lay K, Taieb C, Matucci-Cerinic M. Prevalence of fibromyalgia: a survey in five European countries. Semin Arthritis Rheum. 2010 Jun;39(6):448-53. doi: 10.1016/j.semarthrit.2008.12.003. Epub 2009 Feb 27. PMID 19250656
- [Background] Pastor Mira MA, Lledo Boyer A, Lopez-Roig S, Pons Calatayud N, Martin-Aragon Gelabert M. [Predictors of healthcare resource use in fibromyalgia]. Psicothema. 2010 Nov;22(4):549-55. Spanish. PMID 21044477
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Granero-Molina J, Aguilera-Manrique G, Quesada-Rubio JM, Moreno-Lorenzo C. Benefits of massage-myofascial release therapy on pain, anxiety, quality of sleep, depression, and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:561753. doi: 10.1155/2011/561753. Epub 2010 Dec 28. PMID 21234327
- [Background] Giamberardino MA, Affaitati G, Fabrizio A, Costantini R. Effects of treatment of myofascial trigger points on the pain of fibromyalgia. Curr Pain Headache Rep. 2011 Oct;15(5):393-9. doi: 10.1007/s11916-011-0205-3. PMID 21541831
- [Background] Affaitati G, Costantini R, Fabrizio A, Lapenna D, Tafuri E, Giamberardino MA. Effects of treatment of peripheral pain generators in fibromyalgia patients. Eur J Pain. 2011 Jan;15(1):61-9. doi: 10.1016/j.ejpain.2010.09.002. PMID 20889359
- [Background] Alonso-Blanco C, Fernandez-de-Las-Penas C, de-la-Llave-Rincon AI, Zarco-Moreno P, Galan-Del-Rio F, Svensson P. Characteristics of referred muscle pain to the head from active trigger points in women with myofascial temporomandibular pain and fibromyalgia syndrome. J Headache Pain. 2012 Nov;13(8):625-37. doi: 10.1007/s10194-012-0477-y. Epub 2012 Aug 31. PMID 22935970
- [Background] Alonso-Blanco C, Fernandez-de-las-Penas C, Morales-Cabezas M, Zarco-Moreno P, Ge HY, Florez-Garcia M. Multiple active myofascial trigger points reproduce the overall spontaneous pain pattern in women with fibromyalgia and are related to widespread mechanical hypersensitivity. Clin J Pain. 2011 Jun;27(5):405-13. doi: 10.1097/AJP.0b013e318210110a. PMID 21368661
- [Background] Ge HY, Nie H, Madeleine P, Danneskiold-Samsoe B, Graven-Nielsen T, Arendt-Nielsen L. Contribution of the local and referred pain from active myofascial trigger points in fibromyalgia syndrome. Pain. 2009 Dec 15;147(1-3):233-40. doi: 10.1016/j.pain.2009.09.019. Epub 2009 Oct 9. PMID 19819074
- [Background] Ge HY, Wang Y, Danneskiold-Samsoe B, Graven-Nielsen T, Arendt-Nielsen L. The predetermined sites of examination for tender points in fibromyalgia syndrome are frequently associated with myofascial trigger points. J Pain. 2010 Jul;11(7):644-51. doi: 10.1016/j.jpain.2009.10.006. Epub 2009 Nov 14. PMID 19914876
- [Background] Ge HY. Prevalence of myofascial trigger points in fibromyalgia: the overlap of two common problems. Curr Pain Headache Rep. 2010 Oct;14(5):339-45. doi: 10.1007/s11916-010-0127-5. PMID 20607459
- [Background] Hannuksela M, Vaananen A. The sauna, skin and skin diseases. Ann Clin Res. 1988;20(4):276-8. PMID 3218900
- [Background] Poulsen EU, Jorgensen JO, Madsen FF, Djurhuus JC. Cortical blood-flow in the porcine kidney. A radioactive microsphere study. Urol Res. 1988;16(5):385-7. doi: 10.1007/BF00256048. PMID 3201653
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Vulfsons S, Ratmansky M, Kalichman L. Trigger point needling: techniques and outcome. Curr Pain Headache Rep. 2012 Oct;16(5):407-12. doi: 10.1007/s11916-012-0279-6. PMID 22610507
- [Background] Lim C, Park Y, Bae Y. The effect of the kinesio taping and spiral taping on menstrual pain and premenstrual syndrome. J Phys Ther Sci. 2013 Jul;25(7):761-4. doi: 10.1589/jpts.25.761. Epub 2013 Aug 20. PMID 24259847
- [Background] Fischer AA. Algometry in the daily practice of pain management. J Back Musculoskelet Rehabil. 1997 Jan 1;8(2):151-63. doi: 10.3233/BMR-1997-8209. PMID 24572755
- [Background] Guermazi M, Ghroubi S, Kassis M, Jaziri O, Keskes H, Kessomtini W, Ben Hammouda I, Elleuch MH. [Validity and reliability of Spinal Mouse to assess lumbar flexion]. Ann Readapt Med Phys. 2006 May;49(4):172-7. doi: 10.1016/j.annrmp.2006.03.001. Epub 2006 Mar 20. French. PMID 16630669
- [Background] Ripani M, Di Cesare A, Giombini A, Agnello L, Fagnani F, Pigozzi F. Spinal curvature: comparison of frontal measurements with the Spinal Mouse and radiographic assessment. J Sports Med Phys Fitness. 2008 Dec;48(4):488-94. PMID 18997653
- [Background] Maarek A. Electro interstitial scan system: assessment of 10 years of research and development. Med Devices (Auckl). 2012;5:23-30. doi: 10.2147/MDER.S29319. Epub 2012 Mar 5. PMID 23166454
- [Background] Alexeev VG, Kuznecova LV. Bioimpedance in monitoring of effects of selective serotonin reuptake inhibitor treatment. Psychol Res Behav Manag. 2011;4:81-6. doi: 10.2147/PRBM.S22925. Epub 2011 Jun 30. PMID 22114538
- [Background] Lewis JE, Tannenbaum SL, Gao J, Melillo AB, Long EG, Alonso Y, Konefal J, Woolger JM, Leonard S, Singh PK, Chen L, Tiozzo E. Comparing the accuracy of ES-BC, EIS-GS, and ES Oxi on body composition, autonomic nervous system activity, and cardiac output to standardized assessments. Med Devices (Auckl). 2011;4:169-77. doi: 10.2147/MDER.S24291. Epub 2011 Sep 16. PMID 22915943
- [Derived] Castro-Sanchez AM, Garcia-Lopez H, Mataran-Penarrocha GA, Fernandez-Sanchez M, Fernandez-Sola C, Granero-Molina J, Aguilar-Ferrandiz ME. Effects of Dry Needling on Spinal Mobility and Trigger Points in Patients with Fibromyalgia Syndrome. Pain Physician. 2017 Feb;20(2):37-52. PMID 28158152